CLINICAL TRIAL: NCT03021369
Title: Vergleich Zweier Thoraxdrainage-Systeme in Der Herzchirurgie
Brief Title: Comparison of Two Different Pleural Drainage Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerckhoff Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medela1
Record Dates: First submitted 2017-01-08; First posted 2017-01-13 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Air Leak From Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pleural drainage system Medela (Active Comparator): These patients receive the digital Medela system
  Interventions: Device: Pleural drainage system
- Pleural drainage system Ocean (Active Comparator): These patients receive the analogue Maquet system
  Interventions: Device: Pleural drainage system

INTERVENTIONS:
Device: Pleural drainage system — Pleural drainage system is connected to the chest tubes after surgery.

SUMMARY:
The digital pleural drainage system Topaz+ by Medela is compared to the analogue system Atrium OCEAN by Maquet in patients undergoing cardiac surgery.

The study is prospectively randomized with an all-comer setup. The patients are randomly selected for one of the systems. The surgery is performed in the standard fashion and chest tubes are placed routinely by the surgeon depending on the type of surgery. A retrosternal 32 French drain is placed in every patient and pericardial and/or pleural drains are optional.

The postoperative course does not vary from the clinical standard and the chest tubes are removed according to institutional standard. The clinical data about fluid amount, time of removal, air leaks, tamponade are routinely collected in a digital patient documentation system.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing cardiac surgery
* capability to give informed consent

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Detection of air leak due to lung leakage or injury during surgery by the pleural drainage system. | Occurrence of air leak is until the drain is removed (usually postoperative day 2 or 3)
  The Thopaz+ system displays the amount of air leak on the screen in ml/min and the Ocean system is a 'wet seal' system, where bubbles in the box might indicate an air leak. If air leak is detected, the train cannot be removed and has to stay until no more air leak is detected. If air leak is unclear, chest x-rays with clamped drains are performed. If an pneumothorax is visible in the x-ray, the drains have to stay, otherwise they can be removed safely. The digital air leak detection and quantification by the Thopaz+ system might help in clearly detecting the air leaks.

SECONDARY OUTCOMES:
Time of chest drain removal | Number of days until the chest drains are removed (usually postoperative day 2 or 3, depending on air leak and amount of fluid).
Fluid amount | Total amount of fluid at the time of chest drain removal (usually postoperative day 2 or 3, depending on air leak and amount of fluid).
Number of patients with pericardial tamponade that has to be treated by puncture or surgically | Occurrence through hospital stay (an average of 1 week).
Number of patients with pleural effusion at discharge echo, without intervention | Occurrence through hospital stay (an average of 1 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Germany